CLINICAL TRIAL: NCT00132925
Title: An Efficacy and Safety Evaluation of Nasacort AQ 110 µg QD Children Ages 2-5 Years With Perennial Allergic Rhinitis
Brief Title: An Efficacy and Safety Evaluation of Nasacort AQ in Children Ages 2-5 Years With Perennial Allergic Rhinitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: XRG5029C_3502
Record Dates: First submitted 2005-08-18; First posted 2005-08-22 (Estimated); Last update posted 2011-01-11 (Estimated); Status verified 2011-01

CONDITIONS: Rhinitis, Allergic, Perennial
Keywords: allergic rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Perennial; Rhinitis, Allergic | interventions — Triamcinolone

INTERVENTIONS:
Drug: Triamcinolone

SUMMARY:
The purposes of this study are:

* To demonstrate the efficacy of once daily administration of Nasacort AQ 110 µg compared with placebo in children 2-5 years of age with perennial allergic rhinitis; and
* To assess the safety of Nasacort AQ 110 µg in children 2-5 years of age.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be male or female children ages 2-5 years with a history of at least 1 year of perennial allergic rhinitis (PAR) with or without seasonal allergic rhinitis (SAR) characterized by nasal stuffiness, nasal discharge, sneezing, nasal itching, and total eye symptoms, and verified by positive skin test or radioallergosorbent test (RAST) to perennial allergen that is present in the subject's environment (documented historical testing performed during the past year will be accepted).
* Subjects (assisted by a parent/guardian/care provider) must meet an aggregate symptom score of at least 18 (out of a possible 36) for nasal stuffiness, nasal discharge and sneezing for both the reflective (previous 24 hours) and instantaneous symptom scores recorded in the morning
* Subjects must not have clinically relevant disease other than allergic rhinitis or have clinically relevant deviations from normal on a physical examination.
* Subjects must not have been recently exposed to rhinitis medications prior to screening
* Subjects must have no history of hypersensitivity to glucocorticoids or to any excipients of the formulation
* Subjects undergoing cosyntropin stimulation test must have a morning (8 AM ± 1 hour) pre-stimulation serum cortisol level ≥ 5 µg/dL and 30 minutes post-stimulation serum cortisol level ≥ 18 µg/dL at screening

Exclusion Criteria:

Subjects presenting with any of the following will not be included in the study:

* Asthma, requiring chronic use of inhaled or systemic corticosteroids in the previous 6 months; upper respiratory tract infection or sinus infection requiring antibiotic therapy within 2 weeks prior to screening or viral upper respiratory tract infection within 7 days of screening.
* Nasal polyps, deviated septum, or nasal/facial anatomic abnormalities that interfere with symptom evaluation and/or use of intranasal corticosteroids
* Treatment with more than 2 courses of systemic corticosteroids (each course not exceeding 14 days) within 1 year of screening
* Use of intranasal or ocular corticosteroids within 2 weeks of screening
* Use of oral, inhaled, or intravenous corticosteroids within 1 month of screening
* Use of intramuscular or intra-articular corticosteroids within 3 months of screening
* Use of high potency dermatological corticosteroids within 1 month of screening
* Use of oral leukotriene modifiers within 1 week of screening
* Use of nasal or oral antihistamines or oral or nasal decongestants within 3 days of screening
* Current or history of cataract or glaucoma
* Treatment with any investigational product or use of an investigational device within 1 month of screening
* Immunotherapy, with the exception of a stable maintenance schedule, for at least 1 month prior to screening
* History of hypersensitivity to glucocorticoids or to any excipients of the formulation
* Subject is the investigator or any sub-investigator, research assistant, pharmacist, study coordinator, or other staff or relative thereof directly involved in the conduct of the protocol.

Any waiver of these inclusion and exclusion criteria must be approved by the investigator and the sponsor on a case-by-case basis prior to enrolling the subject. This must be documented by both the sponsor and the investigator.

No subject will be allowed to enroll in this study more than once.

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 460
Dates: Start 2003-11; Study Completion 2006-02

PRIMARY OUTCOMES:
Double-blind phase: Change from baseline in mean daily instantaneous (immediately prior to dosing) Total Nasal Symptom Score (TNSS) over the 4-week double-blind period
Open-label phase: The efficacy variable is the global evaluation of efficacy as rated by the physician and the subject

SECONDARY OUTCOMES:
Change from baseline: in mean daily reflective (previous 24 hours) TNSS over 4-wk double-blind period
for mean daily instantaneous and reflective TNSS by week
for mean instantaneous and reflective daily scores for nasal stuffiness, nasal discharge, sneezing, nasal itching, and total eye symptoms by week and over four week double-blind period

CONTACTS AND LOCATIONS:
Overall Officials: Phyllis Diener, BS, MT (ASCP), Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Inc., Bridgewater, New Jersey, United States

REFERENCES:
- [Derived] Weinstein S, Qaqundah P, Georges G, Nayak A. Efficacy and safety of triamcinolone acetonide aqueous nasal spray in children aged 2 to 5 years with perennial allergic rhinitis: a randomized, double-blind, placebo-controlled study with an open-label extension. Ann Allergy Asthma Immunol. 2009 Apr;102(4):339-47. doi: 10.1016/S1081-1206(10)60340-7. PMID 19441606